CLINICAL TRIAL: NCT01497275
Title: A Phase II Study Evaluating Combined Zevalin(Ibritumomab Tiuxetan)and Velcade(Bortezomib)in Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Zevalin and Velcade in Relapsed/Refractory Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual due to the approval of new drugs for use in Mantle cell lymphoma.
Sponsor: Duke University (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032517
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Mantle-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Bortezomib; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zevalin + Velcade (Experimental): Drug: Rituximab, Bortezomib,Y90 ibritumomab tiuxetan
  Other Names:
  Rituxan Velcade Zevalin
  Rituximab 250mg/m2 will be given on day 1 and on day 8. Bortezomib 1.5mg/m2 will be given on Days 1, 4, 8, and 11. Y90 ibritumomab tiuxetan will be given on Day 8. Dosage will be based on the platelet count obtained at the time of study enrollment. The dose will be 0.4 millicurie (mCi)/kg unless the enrollee's platelets are between 100,000 and 150,000 in which case a dose of 0.3mCi/Kg will be used. Patients who weigh over 80 Kg will receive a maximum dose of 32mCi.
  Interventions: Drug: Rituximab, Bortezomib,Y90 ibritumomab tiuxetan

INTERVENTIONS:
Drug: Rituximab, Bortezomib,Y90 ibritumomab tiuxetan — Rituximab 250mg/m2 will be given on day 1 and on day 8. Bortezomib 1.5mg/m2 will be given on Days 1, 4, 8, and 11. Y90 ibritumomab tiuxetan will be given on Day 8. Dosage will be based on the platelet count obtained at the time of study enrollment. The dose will be 0.4mCi/kg unless the enrollee's platelets are between 100,000 and 150,000 in which case a dose of 0.3mCi/Kg will be used. Patients who weigh over 80 Kg will receive a maximum dose of 32mCi.
  Other Names: Rituxan; Velcade; Zevalin

SUMMARY:
The purpose of this study is to evaluate the effects (good and bad) of the combination of ibritumomab tiuxetan (Zevalin) and bortezomib (Velcade) in patients with relapsed/refractory mantle cell lymphoma.

Zevalin is a monoclonal antibody that is combined with a radioactive substance and given with another monoclonal antibody called rituximab (Rituxan). It works by attaching to cancer cells and releasing radiation to damage those cells. Both Zevalin and Rituxan are given in this study, along with Velcade.

DETAILED DESCRIPTION:
This is a non-randomized, unblinded single arm Phase II trial to evaluate the combination of yttrium90 ibritumomab tiuxetan and bortezomib in patients with relapsed/refractory mantle cell lymphoma (MCL). Standard hematology and chemistries, imaging and bone marrow biopsies will be done.

Research tests: 17cc of blood will be collected at screen, Day 8 OR 11 and month 3. Samples will be collected and stored for future analysis. These analyses may include but are not limited to measurements of proteasome inhibition. No genetic studies will be performed on these samples. Samples will be destroyed at the end of the study.

Primary Objective Estimate the overall response rate (CR + PR) of the combination of bortezomib and ibritumomab tiuxetan in patients with relapsed/refractory mantle cell lymphoma.

Secondary Objectives

* Estimate the progression free and overall survival in patients with relapsed/refractory mantle cell lymphoma who receive bortezomib and ibritumomab tiuxetan.
* Assess the toxicity of the combination of bortezomib and ibritumomab tiuxetan in patients with relapsed/refractory MCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory Mantle Cell lymphoma with measurable disease.
* Age > 18 years old
* Expected survival >/= 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 at initiation of study (Appendix I).
* Laboratory tests meet the levels specified in the protocol

Exclusion Criteria:

* Patients must not have received chemotherapy, radiation or surgical resection of malignancy within 3 weeks of study initiation. However, if they have received nitrosurea or mitomycin C then they should not be enrolled in the study until 6 weeks after therapy was last received.
* No limitations to number of prior therapies
* No prior radioimmunotherapy (RIT)
* Prior bortezomib is allowed
* Patient must be fully recovered from all toxicities associated with prior surgery, radiation treatment, chemotherapy or immunotherapy.
* No active, serious infection or medical or psychiatric illness likely to interfere with participation in this clinic trial
* No known HIV infection
* No active central nervous system (CNS) involvement
* Bone Marrow Involvement >/= 25% within 30 days of initiation of study treatment
* Pregnant or breast feeding
* No patients who have received Granulocyte colony-stimulating factor (G-CSF) or Granulocyte macrophage colony-stimulating factor (GM-CSF) within the 14 days prior to initiating protocol
* No patient who has had major surgery within the four weeks prior to initiating protocol therapy
* No patients with pleural effusion or significant ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Beaven, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started April, 2012 and closed to accrual May, 2014. Patients were recruited from the Cellular Therapy clinic at Duke.
Groups:
- Zevalin + Velcade: Drug: Rituximab, Bortezomib,Y90 ibritumomab tiuxetan Rituximab 250mg/m2 will be given on day 1 and on day 8. Bortezomib 1.5mg/m2 will be given on Days 1, 4, 8, and 11. Y90 ibritumomab tiuxetan will be given on Day 8. Dosage will be based on the platelet count obtained at the time of study enrollment. The dose will be 0.4 millicurie (mCi)/kg unless the enrollee's platelets are between 100,000 and 150,000 in which case a dose of 0.3mCi/Kg will be used. Patients who weigh over 80 Kg will receive a maximum dose of 32mCi.
Period: Overall Study
Arm/Group | Zevalin + Velcade
Started | 5
Completed | 3
Not Completed | 2
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zevalin + Velcade
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  18-49 Years | 1
  50-59 Years | 1
  60-69 Years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response + Partial Response)
Description: Disease will be assessed every 3 months.
  The Cheson criteria will be used to define response:
  Complete Response = Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present prior to therapy.
  Partial Response = A decrease of ≥ 50% in the sum of the products of their greatest transverse diameters (SPD) of up to six of the largest dominant nodes or nodal masses. These nodes or masses should be selected according to the following features: a) they should be clearly measurable in at least two perpendicular measurements; b) they should be from as disparate regions of the body as possible; and c) they should include mediastinal and retroperitoneal areas of disease whenever these sites are involved.
Time Frame: 3 months
Population: Only 3 subjects completed the drug regimen; 1 subject did not complete due to disease progression; 1 did not complete due to adverse event.
Measure: Number; unit: participants
Arm/Group | Zevalin + Velcade
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: Number of Participants With Progression Free Survival
Description: Progression-free survival will be defined as time from on-study to disease progression or death, whichever comes first
Time Frame: 6 months
Population: Only 3 subjects provided evaluable data at the 6 month time point. 2 subjects did not reach this time-point so they were not assessed for progression
Measure: Number; unit: participants
Arm/Group | Zevalin + Velcade
Number analyzed (Participants) | 3
participants | 0

3. Secondary Outcome: Overall Survival at 1 Year
Description: Number of participants who were alive at the 1 year time point. (Overall survival will be defined as the time from on-study to death due to any cause.)
Time Frame: 1 year
Population: 1 subject did not reach the one year evaluation because the study was terminated.
Measure: Number; unit: participants
Arm/Group | Zevalin + Velcade
Number analyzed (Participants) | 4
participants | 2

4. Secondary Outcome: Overall Survival at 5 Year
Description: Number of participants who were alive at the 5 year time point. (Overall survival will be defined as the time from on-study to death due to any cause.)
Time Frame: 5 year
Population: No analysis completed due to study being terminated prior to the 5 year time point.
Arm/Group | Zevalin + Velcade
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Zevalin + Velcade
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin + Velcade (N=5)
other-death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin + Velcade (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Edema-limbs (General disorders) | 1 (1)
Edema-trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
other-herpes zoster (Infections and infestations) | 1 (1)
creatinine increase (Investigations) | 1 (1)
neutrophil count decreased (Investigations) | 1 (1)
platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in extreminity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
rash acne (Skin and subcutaneous tissue disorders) | 1 (1)
thromboembolic event (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed to enrollment due to the approval of new drugs for use in Mantle Cell Lymphoma. We were not able to enroll enough subjects to answer our study questions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes